CLINICAL TRIAL: NCT02425761
Title: A Randomized Controlled Trial of Anterior Versus Posterior Entry Site for Cerebrospinal Fluid Shunt Insertion
Brief Title: The CSF Shunt Entry Site Trial
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Baylor College of Medicine (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); University of Alabama at Birmingham (Other); University of British Columbia (Other); University of Pittsburgh (Other); University of Toronto (Other); University of Utah (Other); University of Washington (Other); Vanderbilt University (Other); Washington University School of Medicine (Other); Hydrocephalus Association (Other); Ohio State University (Other); Johns Hopkins University (Other); University of Calgary (Other); University of Colorado, Denver (Other); University of Southern California (Other)
Responsible Party: Principal Investigator, William Whitehead, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-35639
Record Dates: First submitted 2015-04-20; First posted 2015-04-24 (Estimated); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Hydrocephalus
Keywords: Cerebrospinal Fluid Shunts; Randomized Controlled Trial
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Intervention Model Description: 1 to 1 randomized trial comparing two commonly used shunt insertion entry sites.
Who Masked: Outcomes Assessor
Masking Description: Adjudication committee reviews blinded notes, data collection forms, and films to determine shunt failure.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anterior Entry SIte (Active Comparator): Anterior entry site is defined as shunt surgery with catheter entry into the brain from an opening near the coronal suture, on the top of the head and near the front. Specifically, anterior entry is defined as ventricular catheter entry less than 1 centimeter anterior to the coronal suture near the mid-pupillary line.
  Subjects randomized to this arm will undergo ventriculoperitoneal shunt insertion surgery using an anterior entry site.
  Interventions: Procedure: Ventriculoperitoneal shunt insertion surgery
- Posterior Entry Site (Active Comparator): Posterior entry site is defined as shunt surgery with catheter entry into the brain from an opening near the lambdoid suture, on the back of the head. Specifically, posterior entry is defined as ventricular catheter entry 4 to 7 centimeters above the external occipital protuberance (inion), near the mid-pupillary line.
  Subjects randomized to this arm will undergo ventriculoperitoneal shunt insertion surgery using a posterior entry site.
  Interventions: Procedure: Ventriculoperitoneal shunt insertion surgery

INTERVENTIONS:
Procedure: Ventriculoperitoneal shunt insertion surgery — The most common treatment for hydrocephalus is the placement of a ventriculoperitoneal shunt in the operating room. A shunt is a flexible tube placed into the ventricular system, fluid filled chambers, of the brain that diverts the flow of CSF into another region of the body, usually the abdomen, also known as the peritoneal cavity, where it can be absorbed.

SUMMARY:
The purpose of the study is to compare the survival time (time to first shunt failure) of ventriculoperitoneal (VP) shunts inserted through an anterior entry site with those inserted through a posterior entry site in children. Shunt entry site is the location on the head that the shunt catheter enters the brain on its path to the fluid-filled spaces in the brain, the ventricles. Entry sites can be anterior or posterior.

DETAILED DESCRIPTION:
The study is a multi-centered, randomized, controlled trial comparing two commonly used CSF shunt insertion techniques, anterior and posterior entry site. There is conflicting information and opinions in the pediatric hydrocephalus literature regarding entry site's effect on shunt survival. This trial is designed to detect a 10% or more difference in the rate of shunt survival at one year between the two techniques.

The trial will be conducted by the Hydrocephalus Clinical Research Network and the Hydrocephalus Association. It is a four year study with an estimated sample size of 448 patients. Patients will be randomized in the operating room. Subjects will be followed for a minimum of 18 months.

ELIGIBILITY:
Inclusion Criteria:

1. Less than 18 years of age at the time of shunt insertion; AND
2. Clinical evidence of hydrocephalus that requires a simple ventriculoperitoneal shunt as determined by a pediatric neurosurgeon; AND
3. No prior history of shunt insertion (a history of an external ventricular drain, ventricular reservoir, subgaleal shunt, and or endoscopic third ventriculostomy with or without choroid plexus coagulation is permissible); AND
4. Ventriculomegaly on imaging.

Exclusion Criteria:

1. Need of a shunt that is not a simple ventriculoperitoneal shunt. For example: Patients who require more than one intracranial catheter are excluded. Patients who require a ventricular shunt that terminates in the atrium of the heart, the pleural cavity, the gallbladder, or any other terminal location that is not the peritoneal cavity are excluded. Patients who require a subdural to peritoneal or a cyst to peritoneal shunt are excluded.
2. Active CSF or abdominal infection;
3. CSF leak without hydrocephalus;
4. Pseudotumor cerebri;
5. Hydranencephaly;
6. Loculations within the ventricular system (e.g. large intraventricular cysts or ventricular adhesions which create compartments that distort the ventricular anatomy; isolated trapped lateral ventricle). A small cyst within the ventricle does not meet these criteria;
7. Other difficulties that would preclude follow up at one year (e.g. terminal illness with life expectancy less than 18 months; family plans to move out of region or country);
8. A bilateral scalp, bone, or ventricular lesion that makes placement of either an anterior or a posterior shunt impracticable (e.g. cutis aplasia);
9. Bilateral slit like frontal horns or trigones defined as the widest distance between the medial and lateral walls less than 3 millimeters.
10. Patient is scheduled to have an intra-ventricular procedure (e.g. ETV, endoscopic biopsy, arachnoid cyst fenestration, fenestration of septum pellucidum) in addition to possible or definite VP shunt.

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 448 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Shunt Failure determined by clinical and radiographic findings | Within 18 months to 44 months from shunt insertion surgery
  Shunt failure occurs when the shunt is obstructed, infected, over-drains, or does not drain the entire ventricular system. Shunt failure will be confirmed by radiographic and/ or operative findings, and all failures will be reviewed by a blinded adjudication committee. Subjects will be monitored for shunt failure at each scheduled and unscheduled clinical visit throughout the study. Survival analysis will be used to compare time to shunt failure in each treatment group. The last subject entered into the trial will be followed for 18 months and accrual is expected to take 26 months (maximum follow up 44 months).

SECONDARY OUTCOMES:
Patient quality of life measured by the Pediatric Quality of Life Inventory (PedsQL) | 1 week and 1 year after shunt surgery
  A validated quality of life measure will be administered to all subjects/ caretakers at enrollment and at the above time intervals.
Duration of surgery (minutes) | Shunt insertion surgery
Location of ventricular catheter tip on brain imaging | within 1 year of shunt surgery
  Position of the ventricular catheter on the first postoperative imaging study will be assessed on postoperative imaging studies obtained within 1 year of shunt insertion surgery. The frequency of catheter tips in poor locations (e.g. within brain parenchyma) will be compared between treatment groups.
Number and type of shunt revisions | Within 18 months to 44 months from shunt insertion surgery
  The number of shunt revisions required by each subject from the time of shunt insertion to the conclusion of the study will be compared. All subjects will be followed for at least 18 months.

CONTACTS AND LOCATIONS:
Overall Officials: William E Whitehead, MD, Principal Investigator — Baylor College of Medicine; John Kestle, MD, Study Chair — University of Utah
Locations (14):
- United States (11):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Children's Hospital Colorado, Denver, Colorado
  - Johns Hopkins Children's Center, Baltimore, Maryland
  - St. Louis Children's Hospital, St Louis, Missouri
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Monroe Carell Jr Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Texas Children's Hospital, Houston, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- Canada (3):
  - Alberta Children's Hospital, Calgary, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - The Hospital for Sick Children, Toronto, Ontario

REFERENCES:
- See also: Hydrocephalus Clinical Research Network Website — http://www.hcrn.org
- See also: Hydrocephalus Association Website — http://www.hydroassoc.org/